CLINICAL TRIAL: NCT04313543
Title: Determination of Glycemic Index of Longan Syrup in Healthy Volunteers
Brief Title: Glycemic Index of Longan Syrup in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 827/62
Record Dates: First submitted 2020-03-13; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: Longan; Glycemic; Glucose
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucose and Longan syrup (Experimental): Volunteers take 50 g of glucose in 250 ml of water in 5 minutes.Then, they are tested blood glucose levels (taken from the fingertips) at 15, 30 ,45, 60, 90, and 120 minutes. There is 3 days for wash out period. These tests will be repeated for 3 times for baseline glucose calculation. After that, volunteers take 50 g of longan syrup in 250 ml of water in 5 minutes.Then, they are tested blood glucose levels (taken from the fingertips) at 15, 30 ,45, 60, 90, and 120 minutes. Glycemic index of longan syrup is calculated from area under the curved of blood glucose after longan syrup taking divided to mean of area under the curved of blood glucose after glucose taking
  Interventions: Dietary Supplement: Glucose and Longan syrup

INTERVENTIONS:
Dietary Supplement: Glucose and Longan syrup — Volunteers take 50 g of glucose in 250 ml of water in 5 minutes. Then, they take 50g of longan syrup in 250 ml of water in 5 minutes

SUMMARY:
Volunteers take 50 g of glucose in 250 ml of water in 5 minutes.Then, they are tested blood glucose levels (taken from the fingertips) at 15, 30 ,45, 60, 90, and 120 minutes. There is 3 days for wash out period. These tests will be repeated for 3 times for baseline glucose calculation. After that, volunteers take 50 g of longan syrup in 250 ml of water in 5 minutes.Then, they are tested blood glucose levels (taken from the fingertips) at 15, 30 ,45, 60, 90, and 120 minutes. Glycemic index of longan syrup is calculated from area under the curved of blood glucose after longan syrup taking divided to mean of area under the curved of blood glucose after glucose taking.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-60 years
* Never diagnosis as diabetes mellitus of thyroid dysfunction
* Fasting plasma glucose less than 100 mg/dl
* Body mass index 18.5-24.9 kg/m2
* Be willing to be subjects in this study

Exclusion Criteria:

* Know longan allergy or have history of adverse events from longan
* Take medicines, herbs, or food supplements including thiazide diuretics, beta-blockers ,and estrogen that have an effect on blood sugar level in 1 month before this study starting
* Severe comorbidity or uncontrolled diseases
* Pregnancy and lactation
* Participated in other studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-24 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-03 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | Change from glucose baseline in 120 minutes
  They are tested blood glucose levels (taken from the fingertips) at 15, 30 ,45, 60, 90, and 120 minutes. There is 3 days for wash out period. These tests will be repeated for 3 times for baseline glucose calculation.

SECONDARY OUTCOMES:
Adverse events | 12 days
  Number of participants with skin, respiratory, and gastrointestinal side effects